CLINICAL TRIAL: NCT06741189
Title: Cardiopediatric Home Monitoring Tool
Acronym: OSCAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC24_0146
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Congenital Heart Defect
Keywords: Congenital heart defects, cardiac surgery, care pathway, home monitoring, morbidity and mortality
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard group (Active Comparator): The usual medical monitoring for the first six months postoperatively is standardized between the 4 university hospital centres concerned and consists of :
  1. during the first 4 weeks: a weekly consultation including a record of intercurrent events (malaise, cyanosis, hyperthermia, eating difficulties), a record of weight and vital constants (oxygen saturation, heart rate), an examination of the sternotomy or thoracotomy scar, a clinical cardiovascular examination, a 12-lead electrocardiogram and a transthoracic echocardiogram.
  2. during the following 20 weeks: a consultation at 1, 3 and 6 months including the same assessment procedures.
  Interventions: Other: usual medical monitoring
- home monitoring group (Experimental): In addition to the usual post-operative monitoring, OSCAR home monitoring will enable key parameters to be transmitted to the medical team at a discontinuous rate (once a day for 4 weeks, then once a week for 20 weeks) via a brief questionnaire (smartphone application) and measurement sensors (weight, oxygen saturation, heart rate) linked to an interface, from the first day the patient returns home until the 6th month post-operatively. The values entered will be automatically compared with individualized standards established for each child at a multidisciplinary meeting, and any deviation from the standard will generate an alert. and the response of the medical teams will be protocolized.
  Interventions: Other: Home monitoring; Other: usual medical monitoring

INTERVENTIONS:
Other: Home monitoring — The key parameters (heart rate, arterial oxygen saturation, weight) will be measured at home using the measurement tools used by the parents, and tele-transmitted at a discontinuous rate, i.e. once a day for 4 weeks, then once a week for 20 weeks. The measurement tools will be given to the family before discharge from the hospital ward. These parameters will be entered into the Exolis platform, in addition to a very brief questionnaire designed to provide information about the child's diet, muscle tone and any medication he or she is taking. taken by the child.
  An alert will be automatically generated for the pediatric cardiology team if the data transmitted by the measurement sensors deviates from an individualized standard, defined for each child and/or each care pathway at the multidisciplinary consultation meeting before the child returns home.
  The response will be standardized on the basis of a protocol shared by the 4 investigating centers.
  Arms: home monitoring group
Other: usual medical monitoring — During the first 4 weeks: a weekly consultation including a record of intercurrent events (malaise, cyanosis, hyperthermia, eating difficulties), a record of weight and vital constants (oxygen saturation, heart rate), an examination of the sternotomy or thoracotomy scar, a clinical cardiovascular examination, a 12-lead electrocardiogram and a transthoracic echocardiogram.
  During the following 20 weeks: a consultation at 1, 3 and 6 months including the same assessment procedures.

SUMMARY:
We hypothesize that a home monitoring program combined with routine postoperative care significantly reduces morbidity and mortality after neonatal and pediatric cardiac surgery. This project differs from the previously published experiences by (a) providing an innovative telemedicine solution via the use of validated measurement sensors, (b) an alert system based on individualized standards, established for each care pathway, and (c) a protocolized response from medical teams in the management of alerts generated by the home monitoring tool.

DETAILED DESCRIPTION:
Affecting 12-million people worldwide and 7,400 newborns/year in France, congenital heart defects (CHD) are the leading cause of birth defects and a major cause of morbidity and mortality in childhood.

It is (a) a growing patient population, due to an increase in birth prevalence and survival, and (b) a major public health issue, due to a substantial use of healthcare resources and a dramatic impact on quality of life. CHDs concerned by the OSCAR project are rare diseases (prevalence <1/2000 births) operated on at birth or in infancy. These CHDs expose affected newborns/infants to the risk of major cardiovascular events (fainting, cyanosis, arrhythmias) and/or rapid cardiac decompensation occurring at home in the postoperative period, justifying close ambulatory monitoring to detect early warning signs of complication or decompensation (such as oxygen desaturation, accelerated heart rate, poor weight gain, altered tone, etc.)

This risk is particularly high in certain critical postoperative situations, such as when the physiology of a single ventricle is palliated by a shunt (modified Blalock-Taussig systemic-pulmonary anatomy), or in the intermediate period (interstage) between two palliative surgeries in a Norwood program. In view of the high ambulatory mortality (12-20% in current series) during the interstage of a Norwood program, some expert centers around the world have opted not to discharge operated neonates home, preferring to keep in-hospital monitoring during 4 to 5 months, until stage 2, thus reducing mortality during this critical period. In Anglo-Saxon countries, an outpatient monitoring program has been developed as an alternative for these vulnerable patients, sometimes accompanied by a telemedicine solution, greatly reducing postoperative mortality. This type of outpatient follow-up program does not exist in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 0 and 36 months inclusive
* With a congenital heart defect
* Underwent cardiac surgery at Nantes University Hospital
* Affiliated to a social security scheme
* Free, informed and written consent of the 2 holders of parental authority

Non Inclusion Criteria:

* Clinical or family situation contraindicating a return home
* Physical inability to connect to the Exolis platform at home
* Insufficient understanding on the part of those with parental authority
* Extracardiac co-morbidities responsible for organ failure requiring repeated
* Hospitalisation for non-cardiovascular reasons (e.g. severe renal failure, neurological neurological deficit, complex immune deficiency, etc).
* Patient and/or parents under legal protection

Ages: 0 Minutes to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Estimated)
Dates: Start 2025-09-11 (Estimated); Primary Completion 2027-12-11 (Estimated); Study Completion 2027-12-11 (Estimated)

PRIMARY OUTCOMES:
Reducing postoperative morbidity and mortality | 6th month post-op
  The main objective is to evaluate the impact of home monitoring in reducing postoperative morbidity and mortality in patients aged 0 to 36 months who have undergone MCC.

SECONDARY OUTCOMES:
Children's quality of life | 0,1 month, 3 months and 6 months post op
  Assess the impact of OSCAR surveillance by comparing the 2 groups:
  Children's quality of life during the postoperative period.
Parents' quality of life | 0,1 month, 3 months and 6 months post op
  Assess the impact of OSCAR surveillance by comparing the 2 groups:
  Parents' quality of life during the postoperative period
Parental stress | 0,1 month, 3 months and 6 months post op
  Assess the impact of OSCAR surveillance by comparing the 2 groups:
  Parental stress and family impact during the postoperative period
Children's weight growth | 1 month, 3 months and 6 months post op
  Assess the impact of OSCAR surveillance by comparing the 2 groups:
  Children's weight growth during the postoperative period
Post-traumatic stress syndromes | 6 months post op
  Assess the impact of OSCAR surveillance by comparing the 2 groups:
  The prevalence of post-traumatic stress syndromes in parents at the postoperative month.
Serious non-cardiovascular events | 6 months post op
  Assess the impact of OSCAR surveillance by comparing the 2 groups:
  The rate of serious non-cardiovascular events (in order to study a potential delay in the management of these events in the group with OSCAR monitoring group due to increased follow-up).
Factors other than management | 6 months post op
  To study the impact of factors other than management (OSCAR monitoring versus management) on the parents' quality of life, parental stress and family impact family impact, children's weight gain, and the presence of post-traumatic stress post-traumatic stress disorder in the parents 6 months after the operation.
Therapeutic education program | 6 months post op
  Evaluate the conditions for implementing OSCAR surveillance by assessing :
  The relevance of the OSCAR therapeutic education program (ETP) for the parents in the group concerned.
Acceptability of monitoring for the parents | 6 months post op
  Evaluate the conditions for implementing OSCAR surveillance by assessing :
  The acceptability of monitoring for the parents in the group concerned.
Acceptability of the monitoring for the medical teams | 6 months post op
  Evaluate the conditions for implementing OSCAR surveillance by assessing :
  The acceptability of the monitoring for the medical teams (investigating hospital investigating hospital medical teams and the child's routine care medical teams).
Efficiency | 6 months post op
  Evaluate the conditions for implementing OSCAR surveillance by assessing : its efficiency.

IPD SHARING:
Plan to Share IPD: Undecided